CLINICAL TRIAL: NCT05504343
Title: Assessing The Visual Performance Of Hanita Lenses "Intensity SL" Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanita Lenses (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTF-PM
Record Dates: First submitted 2022-08-01; First posted 2022-08-17 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: single arm single center, open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): This study is a prospective, single arm single center, open label study.
  Interventions: Device: "Intensity SL" Intraocular Lens

INTERVENTIONS:
Device: "Intensity SL" Intraocular Lens — Cataract surgery and intraocular lens implantation

SUMMARY:
The Hanita Lenses Intensity SL IOL is intended for implantation in the capsular bag in the posterior chamber in order to replace the crystalline lens of the eye to attain visual correction of aphakia in adult patients in whom a cataractous lens has been removed, who desire improved uncorrected vision, useful near, intermediate and far visual functions, and reduced spectacle dependence.

DETAILED DESCRIPTION:
Different multifocal intraocular lens (MIOL) designs have been used for more than 25 years1. Unlike conventional mono focal intraocular lenses (IOLs), which bend light to a single focus point on the retina, MIOLs are designed to help patients to see at varying distances using different points of focus2. MIOLs used in clinical practice were either refractive initially, or later diffractive in their optical design. Refractive MIOLs incorporate a lens optic with different optical powers in different parts of the lens, while diffractive MIOLs use diffractive steps on the lens to distribute light rays into two or more principal foci. Irrespective of the design type, however, all MIOLs involve some form of optical compromise and a process of neuroadaptation for the patient3.

Intensity SL intraocular lenses (IOLs) represent the latest in premium lens technology. Intensity SL lenses provide clear vision at all distances - from near to far - thus offering the best chance of true spectacle independence.

Despite the promising results obtained with the latest generation of MIOLs, many surgeons remain reluctant to implant these lenses. Visual symptoms such as glare and haloes, reduced contrast sensitivity and night vision problems are all known complications of multifocal implants and have served to hamper wider acceptance of these IOLs4.

Hanita Lenses new Intensity SL IOL has been designed to have very high efficiency of light leading to a high MTF, wide focal ranges of far, intermediate and near vision and minimal loss of light energy. The main purpose of this study is to evaluate visual acuity and contrast sensitivity patients receiving the new Intensity SL IOL.

ELIGIBILITY:
Inclusion Criteria:

* • Age over 45 years and under 75 years.

  * Patients with bilateral age related cataracts, require bilateral cataract phacoemulsification combined Intraocular Lens implantation;
  * Calculated IOL power is within range 15-30 Diopter (approximate range of axial lengths: 21-25.5mm)
  * Normal corneas with corneal astigmatism below following value:

    1. 1 D if with-the-rule (steep axis is vertical, between 60-120⁰)
    2. 0.4 D if against-the-rule (steep axis is horizontal, 0-30⁰ or 150-180⁰)
    3. 0.7 D if oblique (not one of the cases above)
  * Post-operative best corrected visual acuity expected to be 0.3 logMAR or better.
  * Patient motivated for Intensity SL IOL after screening by surgeon.
  * Fundus visualization is possible.
  * Absence of retinal or optic nerve diseases
  * Signed informed consent

Exclusion Criteria:

* Any of the following condition will render a subject ineligible for inclusion in the analysis:

  * Previous ocular/corneal surgery that may affect refraction accuracy or visual acuity.
  * Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
  * History or evidence of any ocular disease that may affect visual acuity (i.e. uncontrolled glaucoma, ocular injury, corneal pathologies, retinal pathologies in general and macular pathologies in particular, diabetic retinopathy, uveitis, aniridia or iris atrophy, vitreous pathologies (patients with vitreous separation or floaters can be included).
  * Rubella cataract.
  * Amblyopia
  * Significantly dry eye
  * Any other ocular condition that may predispose a subject to future complications or contraindicate implantation of the Intensity SL lens.
  * Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 3.5 mm under mesopic/scotopic conditions)
  * Patients with pupil diameter greater than 4mm in photopic conditions.
  * Pregnant, lactating, or planning to become pregnant during the course of the trial.
  * Allergy or intolerance to required study medications (including antibiotic).
  * Subjects participating in a concurrent clinical trial or if they have participated in an ophthalmology clinical trial within the last 30 days.
  * Traumatic cataract.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Binocular Visual Acuity | 3 months
  Binocular visual acuity for far, intermediate and near distance are measured using an ETDRS chart or PV numbers for distance and PV Numbers Near Vision Card (Precision Vision) for near (40cm) and intermediate distances (80cm).
  Visual acuity is measured in photopic conditions.

SECONDARY OUTCOMES:
Defocus Curve | 3 months
  Defocus Curve is measured using ETDRS chart or PV numbers. A loss of ≥ 3 lines (≥ 15 letters) on an ETDRS chart is considered moderate visual loss. A loss of ≥ 6 lines (≥ 30 letters) is considered severe.
  Patient's pupil diameter will be evaluated using a phoropter to create defocus in 0.5D increments, starting from 1D to -4D relative to emmetropia so that the patient will be corrected for far vision.
Contrast Sensitivity | 3 months
  Contrast Sensitivity is measured using a sine wave gratings chart (FACT) at mesopic and photopic conditions.
  Luminance for photopic conditions will be 85cd/m² and 5cd/m² for mesopic conditions. The working interval for photopic conditions is 75-95cd/m² and for mesopic conditions is 5-15cd/m².
  Luminance for photopic and mesopic conditions will be monitored using Illuminance meter and documented.
Patients Satisfaction | 3 months
  Patient Satisfaction is measured using the modified VF-14 questionnaire for quality of life, in addition to satisfaction questionnaire.
  VF-14 stands for Visual Function questionnaire version 14. Function: High score = better Visual Phenomenon: High score = better Satisfaction: Very happy / Happy / Less Happy / Unhappy

OTHER OUTCOMES:
Toxicity after IOL implantation | 3 months
  Occurrence of adverse events associated with treating patients diagnosed with binocular cataract with Intensity SL IOL implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Suvodip Shaw, Study Director — Dr. Agarwal's Eye Hospital Limited; Dr Ashvin Agarwal, Principal Investigator — Dr. Agarwal's Eye Hospital Limited; Priyanka S., Study Chair — Dr. Agarwal's Eye Hospital Limited
Locations (1):
- Agrawal, Chennai, India